CLINICAL TRIAL: NCT03823352
Title: Open-label, Non-randomized, Phase IIa Study to Evaluate Efficacy and Safety/Tolerability Profiles of Antroquinonol in Adult Patients With Relapsed Acute Myeloid Leukemia (AML) or at Initial Diagnosis When no Intensive Treatment is Possible
Brief Title: Evaluate Efficacy and Safety/Tolerability Profiles of Antroquinonol in Acute Myeloid Leukemia (AML) Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHAML-2-001
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — antroquinonol

STUDY DESIGN:
Intervention Model Description: Patients will receive Antroquinonol 200 mg BID on Day 1 for 4 weeks or until transfusion of red blood cell or platelet ≧ 2, unacceptable toxicity, non-compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antroquinonol (Experimental): Patients will receive Antroquinonol 200 mg BID on Day 1 for 4 weeks or until transfusion of red blood cell or platelet ≧ 2, unacceptable toxicity, non-compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first.
  Interventions: Drug: Antroquinonol

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol: 100 mg and corn oil 100 mg encapsulated in a gelatin capsule administered orally. Dose will be selected(200mg TID or 300mg TID with SOC) after phase I, then follow up the best dose for 40 Patients for the efficacy.
  Other Names: Hocena

SUMMARY:
This is a IIa phase IIa open-label, non-randomized clinical trial of Antroquinonol, capsule, 100 mg (Golden Biotechnology Corporation, Taiwan) in patients with AML.

DETAILED DESCRIPTION:
The given pilot clinical trial of a medicinal product for medical use, is held to evaluate preliminary efficacy and safety/tolerability profiles of antroquinonol in adult patients with relapsed AML or at initial diagnosis when no intensive treatment is possible.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed AML after at least 1 chemotherapy regimen or at initial diagnosis when no intensive treatment possible (based on standard criteria).
2. Men and women 18 to 70 years of age.
3. ECOG performance status = 0 or 1.
4. Ability to comply with the study requirements and give written informed consent.
5. Expected survival more than 3 months.
6. Patients with preserved reproductive potential agree to use, with their partner, adequate contraception throughout the study and for 30 days thereafter (contraceptive methods with reliability greater than 90%: cervical caps with spermicide, diaphragms with spermicide, condoms with intravaginal spermicide, non-hormonal intrauterine devices), or true sexual abstinence.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL).
2. Hemoglobin ≤ 7g/dL or platelet ≤ 50,000.
3. Abnormal liver and renal function:

   * Total bilirubin > 2 mg/dL;
   * AST and ALT > 2.5 × ULN;
   * Creatinine > 1.5 × ULN, OR creatinine clearance < 50 mL/min/1.73m2.
4. The subject has not recovered to grade ≤ 1 adverse events due to investigational or chemotherapeutic drugs or stem cell transplantation which were administered > 4 weeks prior to study enrollment.
5. Patient who has had in the past 3 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast.
6. Subjects with any serious active infection (i.e., requiring an intravenous antibiotic, antifungal, or antiviral agent).
7. Subjects with known human immunodeficiency virus, active hepatitis B or C.
8. Subjects who have any other life-threatening illness or organ system dysfunction, which in the opinion of the Investigator, would either compromise subject safety or interfere with the evaluation of the safety of the study drug.
9. Known or suspected substance abuse or alcohol abuse.
10. Patients with history of seizure disorders or central nervous system leukemia.
11. Patients with uncontrolled, intercurrent illness including, but not limited to, symptomatic neurological illness; active, uncontrolled, systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; significant pulmonary disease or hypoxia; or psychiatric illness/social situations that would limit compliance with study requirements.
12. Inability to swallow oral medications or a recent acute gastrointestinal disorder with diarrhea e.g., Crohn's disease, malabsorption, or CTCAE Grade > 2 diarrhea of any etiology at baseline.
13. Prior major surgery or trauma within 28 days prior to first dose of study drug.
14. A positive urine pregnancy test (strip) for female patients of childbearing potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Complete blood count measurements according International Working Group (IWG) response criteria | 2 weeks
  Evaluation of preliminary efficacy profile of antroquinonol in adult patients with relapsed AML or at initial diagnosis when no intensive treatment is possible.

SECONDARY OUTCOMES:
Number of Participants alive at 4weeks | 4 weeks
  patients' situation
Number of Participants alive at 24 weeks | 24 weeks
  patients' situation

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - City Clinical Hospital n.a. S.P.Botkin, Moscow
  - Tula Regional Clinical Hospital, Tula

IPD SHARING:
Plan to Share IPD: No